CLINICAL TRIAL: NCT06051032
Title: Prospective Randomized Comparative Study on the Incidence of Pulmonary Emboembolism (PE) After Endovascular Treatment of Thrombosed Dialysis Arterio Venous Fistulas (AVF): Balloon Thrombectomy Versus Thromboaspiration Systems.
Brief Title: Compative Study of PE in Thrombosed AVF After Balloon Thrombectomy Vs. Thromboaspiration.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Hospital Universitario Doctor Peset (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-803-1
Record Dates: First submitted 2023-07-12; First posted 2023-09-22 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Embolism and Thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with arteriovenous fistula (AVF) thrombosis and eligible for endovascular treatment, based on predefined inclusion and exclusion criteria, will be enrolled in this study. They will be randomly assigned to receive either balloon thrombectomy or thromboaspiration systems.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Balloon thrombectomy (Experimental): Patients diagnosed with arteriovenous fistula (AVF) thrombosis and deemed eligible for endovascular treatment will undergo balloon thrombectomy.
  Interventions: Device: Balloon thrombectomy
- Thromboaspiration system (Experimental): Patients diagnosed with arteriovenous fistula (AVF) thrombosis and deemed eligible for endovascular treatment will undergo the thromboaspiration system.
  Interventions: Device: Thromboaspiration system

INTERVENTIONS:
Device: Balloon thrombectomy — A specialized catheter with an inflatable balloon at the tip is inserted over a guidewire, previously inserted through the sheath, and advanced to the location of the clot within the blood vessel. The catheter is positioned precisely using fluoroscopic guidance or other imaging modalities. Once positioned, the balloon is inflated, creating pressure against the clot and effectively removing or dislodging it from the vessel walls.
  Arms: Balloon thrombectomy
Device: Thromboaspiration system — The thromboaspiration catheter is carefully guided to the site of the clot within the blood vessel. Once positioned, the suction mechanism is activated, creating a vacuum effect. The catheter gently aspirates or suctions the clot, gradually removing it from the vessel walls. The procedure is performed under fluoroscopic guidance or other imaging modalities to ensure accurate placement of the catheter and successful clot aspiration.
  Arms: Thromboaspiration system

SUMMARY:
The goal of this multicentric clinical trial is to compare the incidence of pulmonary thromboembolism (PTE), assessed through AngioCT, in the endovascular treatment of acute thrombosis in native and prosthetic arteriovenous fistulas (AVF). The main questions it aims to answer are:

* What is the difference in the incidence of pulmonary thromboembolism (PTE) assessed by AngioCT in endovascular treatment of acute thrombosis of native and prosthetic arteriovenous fistulas using balloon thrombectomy versus thromboaspiration systems?
* What is the primary patency rate of arteriovenous fistulas treated with balloon thrombectomy versus thromboaspiration systems?
* What is the clinical success rate in the treatment of arteriovenous fistulas using balloon thrombectomy compared to thromboaspiration systems?
* What are the costs associated with the different thrombectomy techniques in the treatment of arteriovenous fistulas?

Participants will be underwent to balloon thrombectomy versus thromboaspiration systems.

Researchers will compare the patients treated with balloon thrombectomy and thromboaspiration systems to see if the incidence of PE is comparable and to evaluate the primary and secondary patency rates of both thrombectomy techniques, the clinical technical success rate, and the costs associated with each technique.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute thrombosis (< 10 days) of native or prosthetic AVF.

Exclusion Criteria:

* Known pulmonary hypertension.
* Severe pulmonary disease.
* Low cardiopulmonary reserve.
* Recent creation of vascular access.
* Known right left shunt.
* Access infection.
* Allergy to iodinated contrast.
* Patients under 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of PTE after thrombectomy of native and prosthetic AVFs. | The presence of PTE will be evaluated within 24 hours after treatment.
  The following parameters will be assessed: Dialysis flow (mL/min), Dialysis Recirculation (%), Dialysis BP (Normal; Elevated), Dialysis PV (Normal; Elevated), Dialysis dose (Kt), Adequate dialysis (Yes, Not), Doppler AVF (Patent; Residual stenosis; Retrombosis; Thrombosis), PET presence (Yes, Not), PET location (Multilobar; Lobar; Segmental; Subsegmental), Hemodynamic overload, Pulmonary artery caliber (mm), Ventricle diameter dx (mm), RV/LV ratio (%), PET effect (Symptomatic; Asymptomatic)
PTE resolution rate 1 month after thrombectomy of native and prosthetic AVFs. | The resolution of PTE will be evaluated 1-month after the treatment
  The following parameters will be assessed: Dialysis flow (mL/min), Dialysis Recirculation (%), Dialysis BP (Normal; Elevated), Dialysis PV (Normal; Elevated), Dialysis dose (Kt), Adequate dialysis (Yes, Not), Doppler AVF (Patent; Residual stenosis; Retrombosis; Thrombosis), PET resolution (Yes, Not), Hemodynamic overload, Pulmonary artery caliber (mm), Ventricle diameter dx (mm), RV/LV ratio (%), PET effect (Symptomatic; Asymptomatic)

CONTACTS AND LOCATIONS:
Overall Officials: José Martínez Rodrigo, Principal Investigator — Hospital Universitario La Fe
Locations (1):
- Hospital La Fe, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Fonseca AV, Toledo Barros MG, Baptista-Silva JC, Amorim JE, Vasconcelos V. Interventions for thrombosed haemodialysis arteriovenous fistulas and grafts. Cochrane Database Syst Rev. 2024 Feb 14;2(2):CD013293. doi: 10.1002/14651858.CD013293.pub2. PMID 38353936